CLINICAL TRIAL: NCT00863460
Title: Prospective , Multicentric, Randomized Phase II Study, Evaluating the Role of Cranial Radiotherapy or Intensive Chemotherapy With Hematopoietic Stem Cell Rescue After Conventional Chemotherapy for Primary Central Nervous System in Young Patients (< 60 y)
Brief Title: Cranial Radiotherapy or Intensive Chemotherapy With Hematopoietic Stem Cell Rescue for Primary Central Nervous System Lymphoma in Young Patients
Acronym: PRECIS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Ministry of Health, France (Other Government); Hoffmann-La Roche (Industry); Amgen (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRH 07/422/H; EudraCT N° 2007-005378-30
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): MTX-based chemotherapy followed by WBRT
  Interventions: Radiation: cranial radiotherapy; Drug: MTX based chemotherapy
- B (Experimental): MTX-based chemotherapy followed by intensive chemotherapy and hematopoietic stem cell rescue
  Interventions: Drug: intensive chemotherapy and hematopoietic stem cell rescue; Drug: MTX based chemotherapy

INTERVENTIONS:
Radiation: cranial radiotherapy — 40 Gy
  Arms: A
Drug: intensive chemotherapy and hematopoietic stem cell rescue — intensive chemotherapy and hematopoietic stem cell rescue
  Other Names: Thiotepa IV (250 mg/m²/day) day-9 day-8 day-7; Busulfan IV (0.8 mg/kg X 10) day-6 to day-4; Cyclophosphamide IV (60 mg/kg/day) day-3 & day-2; Reinjection of hematopoietic stem cells day0
  Arms: B
Drug: MTX based chemotherapy — R-MBVP 2 cycles day1 and day28 followed by R-Aracytine 2 cycles days58&59 and days79&80
  Other Names: R-RMVP :; Rituximab IV if LNH type B (375 mg/m²) day1; Methotrexate IV (3g/m² during 30 minutes) day1 and day15; Etoposide IV (100 mg/m²) day2; Carmustine IV (100 mg/m²) day3; Prednisone PO (60 mg/m²/day)day1 to day5; R-Aracytine :; Aracytine IV (3g/m²) day1 & day2

SUMMARY:
Purpose of the study :

To evaluate the antitumoral effect of two therapeutic procedures and to evaluate their respective toxicity on the CNS.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically proven diagnostic of Primary CNS lymphoma
* All histological types of non-Hodgkin's lymphoma, except MALT
* Age > 18 and < 60 ans.
* Negative for HIV, HCV and HBV
* Written informed consent -

Exclusion Criteria:

* Age < 18 or > 60 ans
* Isolated intra-ocular lymphoma
* Previous history of indolent lymphoma
* Previous chemotherapy or radiotherapy for PCNSL
* Isolated CNS relapse of systemic NHL
* Previous history of cancer in the last 5 years, except basocellular carcinoma and non invasive cervix cancer
* Renal insufficiency or creatinin clearance < 60 ml/min
* Liver enzymes > 3N.
* Platelets < 100 000/mm3 or neutrophils < 1500/mm3)
* Previous history of organ transplantation or other cause of severe immunodeficiency
* Pregnancy or active sexual women with no contraception
* Unable to follow the protocol for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2008-10-03 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
2-years progression-free survival in each arm | 2 years after inclusion

SECONDARY OUTCOMES:
Overall response rate at the end of the procedure | at the end of procedure at 1 and 2 years
Overall survival | 2 years after inclusion
Event-free survival | 2 years after inclusion
Neurotoxicity | each years during ten years

CONTACTS AND LOCATIONS:
Overall Officials: Carole Soussain, MD, Principal Investigator — Institut Curie - Hôpital René Huguenin
Locations (23):
- France (23):
  - Cancérologie Hôpital Sud, Amiens
  - Chu D'Angers, Angers
  - CHR Argenteuil, Argenteuil
  - CHU de Besancon, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Hôtel Dieu, Clermont-Ferrand
  - CHU Michalon, Grenoble
  - Centre Hospitalier Lens, Lens
  - CHU de Limoges, Limoges
  - CHU de la Timone, Marseille
  - Hôtel Dieu Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nimes, Nîmes
  - GH Pitié-Salpétrière, Paris
  - CHG Saint Jean, Perpignan
  - CHU Hôpital Bernard, Poitiers
  - Chu Reims, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie, Saint-Priest-en-Jarez
  - CH de Saint-Quentin, Saint-Quentin
  - Hôpital Bretonneau, Tours
  - CHU Nancy - Hôpital Neurologique, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Houillier C, Dureau S, Taillandier L, Houot R, Chinot O, Molucon-Chabrot C, Schmitt A, Gressin R, Choquet S, Damaj G, Peyrade F, Abraham J, Delwail V, Gyan E, Sanhes L, Cornillon J, Garidi R, Delmer A, Al Jijakli A, Morel P, Waultier A, Paillassa J, Chauchet A, Gastinne T, Laadhari M, Plissonnier AS, Feuvret L, Cassoux N, Touitou V, Ricard D, Hoang-Xuan K, Soussain C; LOC Network for CNS Lymphoma. Radiotherapy or Autologous Stem-Cell Transplantation for Primary CNS Lymphoma in Patients Age 60 Years and Younger: Long-Term Results of the Randomized Phase II PRECIS Study. J Clin Oncol. 2022 Nov 10;40(32):3692-3698. doi: 10.1200/JCO.22.00491. Epub 2022 Jul 14. PMID 35834762
- [Derived] Houillier C, Taillandier L, Dureau S, Lamy T, Laadhari M, Chinot O, Molucon-Chabrot C, Soubeyran P, Gressin R, Choquet S, Damaj G, Thyss A, Abraham J, Delwail V, Gyan E, Sanhes L, Cornillon J, Garidi R, Delmer A, Tanguy ML, Al Jijakli A, Morel P, Bourquard P, Moles MP, Chauchet A, Gastinne T, Constans JM, Langer A, Martin A, Moisson P, Lacomblez L, Martin-Duverneuil N, Delgadillo D, Turbiez I, Feuvret L, Cassoux N, Touitou V, Ricard D, Hoang-Xuan K, Soussain C; Intergroupe GOELAMS-ANOCEF and the LOC Network for CNS Lymphoma. Radiotherapy or Autologous Stem-Cell Transplantation for Primary CNS Lymphoma in Patients 60 Years of Age and Younger: Results of the Intergroup ANOCEF-GOELAMS Randomized Phase II PRECIS Study. J Clin Oncol. 2019 Apr 1;37(10):823-833. doi: 10.1200/JCO.18.00306. Epub 2019 Feb 20. PMID 30785830